CLINICAL TRIAL: NCT05514535
Title: Efficacy and Safety of Once-weekly Semaglutide S.C. 2.0 mg as Add-on to Dose-reduced Insulin Glargine vs Titrated Insulin Glargine in Participants With Type 2 Diabetes and Overweight
Brief Title: A Research Study to Look Into How Semaglutide, Together With a Lower Dose of Insulin Glargine, Compares to a Higher Dose of Insulin Glargine Alone in People With Type 2 Diabetes (SUSTAIN OPTIMIZE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4801; U1111-1267-0312 (Other: World Health Organization (WHO)); 2021-004392-13 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insuline glargine U100 (reduced) + semaglutide (Experimental): Participants will initially receive 0.25 milligrams (mg) once-weekly semaglutide subcutaneously (s.c.) and the dose will be gradually escalated to 2 mg as an add-on to dose-reduced insulin glargine s.c. given once-daily. Insulin glargine U100 will be reduced by 10 U at the initiation of semaglutide and then again at each semaglutide dose escalation. Insulin glargine dose will be adjusted based on the mean of three pre-breakfast self-measured plasma glucose (SMPG) values (target SMPG: 4.4-7.2 millimoles per litre (mmol/L)).
  Interventions: Drug: Semaglutide; Drug: Insuline glargine U100 (reduced)
- Insuline glargine U100 (titrated) (Active Comparator): Participants will receive titrated insuline glargine U100 s.c. once-daily. Insulin glargine U100 dose will be adjusted based on the mean of three pre-breakfast SMPG values (target SMPG: 4.4-7.2 mmol/L).
  Interventions: Drug: Insuline glargine U100 (titrated)

INTERVENTIONS:
Drug: Semaglutide — Participants will receive once-weekly semaglutide s.c. for 40 weeks. Semaglutide 0.25 mg will be given at week 0 and then the dose will be escalated at weeks 4, 8 and 12 to 0.5 mg, 1 mg, 2 mg respectively.
  Arms: Insuline glargine U100 (reduced) + semaglutide
Drug: Insuline glargine U100 (reduced) — Participants will receive insulin glargine U100 s.c. once-daily. Insulin glargine dose will be reduced by 10 U at initiation of semaglutide and then again at each semaglutide dose escalation up to 40 weeks. The dose will be adjusted based on the mean of three pre-breakfast SMPG values (target SMPG: 4.4-7.2 mmol/L).
  Arms: Insuline glargine U100 (reduced) + semaglutide
Drug: Insuline glargine U100 (titrated) — Participants will receive titrated insulin glargine U100 s.c. once-daily up to 40 weeks. The dose will be adjusted based on the mean of three pre-breakfast SMPG values (target SMPG: 4.4-7.2 mmol/L).
  Arms: Insuline glargine U100 (titrated)

SUMMARY:
This study compares semaglutide, together with a lower dose of insulin glargine, to a higher dose of insulin glargine in participants with type 2 diabetes. The study looks at how well the study medicines control blood glucose levels. Participants will either get semaglutide together with a lower dose of insulin glargine or a higher dose of insulin glargine. The study will last for about 47 weeks (approximately 11 months). Participants will have 9 clinic visits, 15 phone/video calls and 1 home visit. Participants will be asked to wear a sensor that measures their blood sugar all the time in 2 periods of 10 days during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2D) mellitus greater than or equal to (>=) 180 days before screening.
* Glycated haemoglobin (HbA1c) of 7-10 percentage [(53-86 millimoles per mole (mmol/mol)] (both inclusive) as assessed by central laboratory on the day of screening.
* Body mass index (BMI) greater than or equal to (>=) 25 kilograms per meter square (kg/m^2) on the day of screening.
* Stable daily dose(s) greater than or equal to (>=) 90 days before screening of any of the following anti-diabetic drugs or combination regimens:
* Any metformin formulations greater than or equal to (>=) 1500 milligrams (mg) or maximum tolerated or effective dose.
* Any metformin combination formulation greater than or equal to (>=) 1500 mg or maximum tolerated or effective dose.

The treatment can be with or without sodium glucose cotransporter 2 (SGLT-2) inhibitors.

• Treated with a once daily basal insulin (e.g. insulin glargine Unit 100 or U300, neutral protamine hagedorn (NPH) insulin, insulin detemir, insulin degludec) less than or equal to (<=) 40 units/day (U/day) for greater than or equal to (>=) 90 days before screening. Short-term bolus insulin treatment for a maximum of 14 days before screening is allowed.

Exclusion Criteria:

* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Potentially missed diagnosis of Type 1 diabetes (T1D) or latent autoimmune diabetes in adults (LADA) verified by C-peptide less than 0.26 nanomoles per litre (nmol/L) (or 260 picomoles per liter [pmol/L] [0.78 nanograms per millilitre {ng/mL}]) or antibodies to glutamic acid decarboxylase (anti-GAD) greater than 5 units/millilitre, as measured by the central laboratory at screening.
* Presence or history of pancreatitis (acute or chronic).
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of less than 30 millilitre per minute per 1.73 meter square at screening as defined by Kidney Disease: Improving Global Outcomes (KDIGO) 2012 classification.
* Any episodes of diabetic ketoacidosis within 90 days before screening.
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question 8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 40)
  Non-inferiority of semaglutide s.c. as add-on to dose-reduced insulin glargine to that of titrated insulin glargine will be assessed based on the clinically acceptable margin of 0.3 percentage (%) for the mean treatment difference in HbA1c. Measured as percentage.

SECONDARY OUTCOMES:
Change in Body Weight | From baseline (week 0) to end of treatment (week 40)
  Measured as kilogram
Relative Change in Daily Insulin Dose | From baseline (week 0) to end of treatment (week 40)
  Measured as percentage
Change in HbA1c | From baseline (week 0) to end of treatment (week 40)
  Superiority of semaglutide s.c. as add-on to dose-reduced insulin glargine versus titrated insulin glargine will be assessed. Measured as percentage.
Score of Diabetes Treatment Satisfaction Questionnaire - Change Version (DTSQc) | At end of treatment (week 40)
  The questionnaire has been designed to measure the change in the level of satisfaction with diabetes treatment regimens in participants with diabetes who have had a recent intervention. It consists of 8 questions, which are to be answered on a Likert scale from -3 to +3 (-3 = much less satisfied now to +3 = much more satisfied now), with 0 (midpoint), representing no change. Six questions are summed to produce a total treatment satisfaction score. The remaining two questions concern perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively. The DTSQc total treatment satisfaction score ranges from -18 to +18, with higher scores associated with greater treatment satisfaction. Measured as score on a scale.
Participants Achieving: Insulin Dose Equal to 0 Units (Yes/No) | At end of treatment (week 40)
  Measured as count of participants
Participants Achieving: Insulin Dose Reduced From Baseline by at Least 50 Percentage (Yes/No) | At end of treatment (week 40)
  Measured as count of participants
Participants Achieving: HbA1c less than 7 Percentage (Yes/No) | At end of treatment (week 40)
  Measured as count of participants
Number of Severe Hypoglycaemic Episodes (Level 3) | From baseline (week 0) to end of treatment (week 40)
  Measured as number of episodes
Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 Millimoles Per Litre (mmol/L) [54 Milligrams Per Decilitre (mg/dL)] Confirmed by Blood Glucose Meter) | From baseline (week 0) to end of treatment (week 40)
  Measured as number of episodes
Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL), Confirmed by Blood Glucose Meter) or Severe Hypoglycaemic Episodes (Level 3) | From baseline (week 0) to end of treatment (week 40)
  Measured as number of episodes
Participants Achieving All of The Following Targets: HbA1c Reduced From Baseline by At Least 0.3 %; Insulin Dose Reduced From Baseline; No Hypoglycaemic Episodes; No Weight Gain | At end of treatment (week 40)
  No hypoglycaemic episodes defined as less than 3.9 mmol/L [70 milligrams per decilitre (mg/dL)] confirmed by Blood Glucose meter. Outcome measure measured as count of participants.
Change in Score of Diabetes Treatment Satisfaction Questionnaire - Status Version (DTSQs) | From baseline (week 0) to end of treatment (week 40)
  The questionnaire has been designed to measure satisfaction with diabetes treatment regimens in participants with diabetes. The questionnaire contains 8 components and measures the treatment for diabetes (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings regarding treatment. The value presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction. Measured as score on a scale.
Change in Score of Short Form 36 Version 2 (SF-36 v2) | From baseline (week 0) to end of treatment (week 40)
  The SF-36 v2 will be used to measure differences in quality of life and mental wellbeing. The scores 0-100 (where higher scores indicated a better quality of life and mental wellbeing) from the SF-36 will be converted to a norm-based score using a T-score transformation in order to obtain a direct interpretation in relation to the distribution of the scores in the 1998 United States general population. Measured as score on a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (153):
- United States (76):
  - Lenzmeier Fam Med CCT Research, Glendale, Arizona
  - San Fernando Valley Hlth Inst, LLC, Canoga Park, California
  - John Muir Physicians Network, Concord, California
  - Valley Research, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - Velocity Clinical Research Huntington Park, Huntington Park, California
  - Velocity Clin Res San Diego, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - Loma Linda Univ Hlth Cr Endo, Loma Linda, California
  - Downtown LA Res Ctr. Inc., Los Angeles, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Wetlin Research Associates, Inc., San Diego, California
  - Encore Medical Research LLC, Hollywood, Florida
  - Northeast Res Inst. Inc., Jacksonville, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - New Horizon Research Center, Miami, Florida
  - Elite Research Center, Miami, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - International Research Associates, LLC_Miami, Miami, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - Suncoast Clinical Research, Inc._New Port Richey, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - CVS Store Number: 7689, Atlanta, Georgia
  - Coastal Heritage Clinical Research, Hinesville, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - CVS Store Number: 05520, Savannah, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Brengle Family Medicine, Indianapolis, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - AMR New Orleans, New Orleans, Louisiana
  - Ileana J. Tandron, MD APMC (a private medical office), Slidell, Louisiana
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - Endo And Metab Cons, Rockville, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - Elite Research Center, Flint, Michigan
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Mercury Str Med Grp, PLLC, Butte, Montana
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - AMC Community Endocrinology, Albany, New York
  - Mid Hudson Med Res-New Windsor, New Windsor, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Lucas Research Inc., Morehead City, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Velocity Clin Res Cleveland, Beachwood, Ohio
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - University of Toledo_Toledo, Toledo, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Accellacare US Inc., d/b/a Accellacare of Knoxville, Knoxville, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Thyroid Endocrinology & Diabetes PA, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - San Antonio Prem Int Med, San Antonio, Texas
  - Diabetes Glandular Diseases Clinic, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Virginia Endo Res, LLC, Chesapeake, Virginia
  - CVS Store Number: 01396, Reston, Virginia
  - CVS Store Number: 1537, Richmond, Virginia
  - Amherst Family Practice P.C., Winchester, Virginia
  - WVU Medicine, Morgantown, West Virginia
- Czechia (6):
  - EDUMED s.r.o., Náchod
  - Diahelp - diabetologie, Pardubice
  - MUDr. Jitka Zemanova - diabetologie a interna, s.r.o., Plzen - Vychodni Predmesti
  - Diabet2 s.r.o., Prague
  - MUDr. Michala Pelikanova, Prague
  - ResTrial s.r.o., Prague
- Greece (10):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - University Hospital of Alexandroupolis, Alexandroupoli
  - "Laiko" General Hospital of Athens, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - General Hospital of Nikaia, Nikaia
  - Tzaneio General Hospital of Piraeus, Piraeus
  - AHEPA General University Hospital, Thessaloniki
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
- Italy (10):
  - A.O.U. Università Studi della Campania "Luigi Vanvitelli", Napoli, Campania
  - Ospedale Santa Maria Goretti - UOD Diabetologia, Latina, LT
  - Azienda Unita' Sanitaria Locale Toscana Nord Ovest - Cittadella della Salute Campo di Marte, Lucca, LU
  - Istituto Scientifico San Raffaele, Milan, MI
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia, Umbria
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Policlinico Mater Domini Università di Catanzaro, Catanzaro
  - ASST degli Spedali Civili di Brescia-Presidio Ospedaliero di Montichiari, Montichiari
  - A.O.U. Università Studi della Campania "Luigi Vanvitelli", Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Dipartimento di scienze Mediche e Chirurgiche, Rome
- Portugal (9):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - Unidade Local De Saude De Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - Unidade Local De Saude Da Regiao De Aveiro E.P.E., Aveiro
  - Unidade de Local de Saúde de Braga, Braga
  - Unidade Local De Saude Do Oeste E.P.E., Caldas da Rainha
  - Unidade Local De Saude Da Regiao De Leiria E.P.E.- Hospital de Santo André, Leiria
  - Unidade Local de Saúde de São José EPE - Hospital Curry Cabral, Lisbon
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital Egas Moniz, Lisbon
  - Unidade Local de Saúde do Alto Minho E.P.E. - Viana do Castelo, Viana do Castelo
- Romania (15):
  - SC Grand Med SRL, Oradea, Bihor County
  - Spitalul Judetean de Urgenta Targoviste, Târgovişte, Dâmbovița County
  - CMI Dr Pop Lavinia, Baia Mare, Maramureş
  - Novus Medical Clinica SRL, Ploieşti, Prahova
  - Centrul Medical Sfantul Stefan, Timișoara, Timiș County
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - Clinica Grivitei 224 S.R.L., Brăila
  - Diabs&Nutricare Srl, Bucharest
  - Clinic of Diabetes Constanta, Constanța
  - Clinical Emergency Sf. Apostol Andrei Hospital, Galati
  - SC Consultmed SRL, Iași
  - Medical Practice SRL, Oradea
  - S.C. Dianutrilife Medica S.R.L., Ploieşti
  - Clinica Korall S.R.L. Satu Mare, Satu Mare
  - Dentosim Queen Srl, Târgu Mureş
- Slovakia (10):
  - DIA - CLARUS s.r.o., Bojnice
  - MediTask, s.r.o, Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava
  - Diabetologicka ambulancia DIA-MAX s.r.o., Levice
  - IN-DIA s.r.o., Lučenec
  - FUNKYSTUFF s.r.o, Nové Zámky
  - Diakom, spol. s r.o., Poprad
  - DIALIPID, s.r.o., Prešov
  - Tatratrial s.r.o., Rožňava
  - BENROD s.r.o., Štúrovo
- South Africa (7):
  - Diabetes Care Centre & CDE Centre, Benoni, Gauteng
  - East Rand Physicians, Benoni, Gauteng
  - East Rand Physicians, Johannesburg, Gauteng
  - Centre for Diabetes, Johannesburg, Gauteng
  - Dr J Reddy, Durban, KwaZulu-Natal
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal
  - Dr T Padayachee, eMkhomazi, KwaZulu-Natal
- Spain (6):
  - Centro Periférico de Especialidades Bola Azul, Almería
  - ABS La Roca del Vallés_Endocrinología, La Roca Del Vallés
  - ABS La Roca del Vallés, La Roca Del Vallés
  - Hospital Infanta Leonor, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Infanta Luisa, Seville
- Ukraine (4):
  - Kharkiv Regional Clinical Hospital - Endocrinology department, Kharkiv
  - Khmelnytskyi Regional Hospital - Endocrinology department, Khmelnytskyi
  - Ternopil Central District Hospital - Outpatient department, Ternopil
  - Medical centre"Elitmedservis"LLC, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com